CLINICAL TRIAL: NCT07087912
Title: Safety and Immunogenicity of the Live Attenuated Tetravalent Butantan-Dengue Vaccine (Butantan-DV) in Patients With Autoimmune Rheumatic Diseases Living in Dengue-Endemic Areas
Brief Title: Safety and Immunogenicity of the Live Attenuated Tetravalent Butantan-Dengue Vaccine in Autoimmune Rheumatic Diseases
Acronym: BTNDV-ARD
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Butantan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 89470625.3.0000.0068
Record Dates: First submitted 2025-06-30; First posted 2025-07-28 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-11

CONDITIONS: Rheumatoid Arthritis (RA); Juvenile Idiopathic Arthritis (JIA); Systemic Lupus Erythematosus (SLE); Juvenile Systemic Lupus Erythematosus; Systemic Sclerosis (SSc); Idiopathic Inflammatory Myopathies (IIMs); Axial Spondyloarthritis; Psoriatic Arthritis (PsA); Granulomatosis With Polyangiitis; Microscopic Polyangiitis; Antiphospholipid Syndrome; Takayasu Arteritis
Keywords: Tetravalent Vaccine; Butantan-Dengue Vaccine; Autoimmune Rheumatic Diseases; Rheumatology; Pediatric Rheumatology; Infectious Disease Prevention; Vaccine
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Juvenile; Lupus Erythematosus, Systemic; Scleroderma, Systemic; Myositis; Axial Spondyloarthritis; Arthritis, Psoriatic; Granulomatosis with Polyangiitis; Microscopic Polyangiitis; Antiphospholipid Syndrome; Takayasu Arteritis | interventions — Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ARDs (Experimental): Patients with ARDs will receive 0.5 mL subcutaneous dose of Butantan-DV
  Interventions: Biological: Dengue 1,2,3,4 (attenuated) vaccine
- Control (Active Comparator): Healthy subjects will receive 0.5 mL subcutaneous dose of Butantan-DV
  Interventions: Biological: Dengue 1,2,3,4 (attenuated) vaccine

INTERVENTIONS:
Biological: Dengue 1,2,3,4 (attenuated) vaccine — A single 0.5 mL dose of the live attenuated tetravalent dengue vaccine (Butantan-DV), administered subcutaneously on Day 1. The vaccine contains attenuated viral strains for DENV-1, DENV-3, DENV-4, and a chimeric DENV-2 component. It is manufactured and formulated by the Instituto Butantan (São Paulo, Brazil).
  Other Names: Butantan-DV; TetraVax-DV-TV003

SUMMARY:
The goal of this clinical trial is to evaluate whether the live attenuated tetravalent Butantan-Dengue vaccine (Butantan-DV) is safe and capable of inducing an immune response in patients aged 12 to 59 years with autoimmune rheumatic diseases (ARDs) who are clinically stable and under low-grade or no immunosuppression, as well as in healthy volunteers matched by sex and age.

The main questions it aims to answer are:

Does the vaccine induce adequate seroconversion in patients with ARDs compared to healthy controls? What is the frequency and intensity of common adverse events after vaccination in ARDs patients? Does physical activity levels and nutritional status influence vaccine-induced immune response in patients with ARDs?

Researchers will compare patients with ARDs to healthy controls to evaluate if the vaccine elicits similar immune responses and safety profiles.

All participants will:

* receive a single 0.5 mL dose of the Butantan-DV vaccine via subcutaneous injection;
* undergo blood sample collection before and after vaccination (baseline, Day 42, and Day 400) to assess antibody and cellular responses;
* attend follow-up visits on Days 7, 14, and 42 for safety monitoring and laboratory tests;
* report any symptoms or adverse events using a standardized diary for 42 days;
* be followed for up to one year for long-term safety and immunogenicity assessments.
* wear a device for 14 consecutive days to assess current and habitual physical activity levels.
* answer three non-consecutive 24-hour dietary recalls, including at least one weekend day to assess nutritional status.
* collect blood samples one-year after vaccination to access immunogenicity and cellular response.

Researcher will also perform subgroups analysis in:

A viremia subgroup (50 patients and 50 healthy controls) will provide additional samples on Days 1, 7, 14, 28, 42, and-if viremia is detected-Day 68, to evaluate post-vaccination viremia and its duration.

An immunogenicity subgroup (~20% of participants, n=96) will undergo cellular immune response testing via flow cytometry to evaluate T-cell responses.

DETAILED DESCRIPTION:
Dengue is hyper-endemic in Brazil, with millions of probable cases and a growing burden of hospitalisation and death each year. Patients with autoimmune rheumatic diseases (ARDs) are especially vulnerable because their underlying immune dysregulation and the use of immunosuppressive agents increase the risk of severe infection and poor outcomes. Current rheumatology guidelines recommend vaccination, yet live-attenuated products are traditionally avoided unless immunosuppression is minimal, leaving an important evidence gap for this population.

The Butantan-DV vaccine is a single-dose, tetravalent, live-attenuated formulation derived from all four dengue serotypes. Phase II-III data in the general population have demonstrated an overall efficacy of ~80 % and an acceptable safety profile, with clear operational advantages over other licensed vaccines (broader age indication and single-dose schedule). However, its immunogenicity and safety have not been prospectively examined in ARD patients under low-grade or no immunosuppression-precisely the subgroup for whom live vaccines may be permissible but still pose theoretical risks.

This open-label, Phase IIIb, prospective study will enrol 318 clinically stable ARD patients (ages 12-59 years) on low-grade or no immunosuppression and 159 age- and sex-matched healthy controls living in dengue-endemic areas. All participants receive a single 0.5 mL subcutaneous dose of Butantan-DV on Day 1. Core follow-up visits occur on Days 7, 14 and 42 for clinical assessment, laboratory safety panels and adverse-event diary review; long-term surveillance continues to Day 400 to characterise antibody persistence and late safety signals.

Two exploratory components will be evaluated:

Viremia substudy: 50 patients and 50 controls undergo additional sampling on Days 1, 7, 14, 28, 42 (and Day 68 if viraemic) to quantify the incidence, magnitude and duration of post-vaccination viremia by multiplex RT-PCR.

Cellular-immunity substudy: ~20 % of participants provide peripheral blood mononuclear cells at baseline, Day 42 and Day 400 for intracellular cytokine staining to define CD8+ T-cell responses against pooled dengue peptides, filling a key knowledge gap on cell-mediated protection in immunocompromised hosts.

Safety oversight is reinforced by a predefined toxicity-grading schema, 24-hour study hotline, systematic capture of solicited/unsolicited adverse events through Day 42, and independent Data and Safety Monitoring Board review at six-month intervals or ad-hoc for any serious events.

Disease-activity flares will be tracked with validated indices tailored to each ARD diagnosis (e.g., DAS-28, SLEDAI-2K, ASDAS) on Days 1 and 42 to distinguish vaccine reactogenicity from underlying disease exacerbation.

Physical activity will be assessed using validated questionnaires at D1 and objective accelerometry (D1-D14), while dietary intake will be evaluated through repeated 24-hour dietary recalls and food quality classification starting at D1.

The primary scientific contribution is to establish whether seroconversion rates (PRNT50) in low-grade immunosuppressed ARD patients are non-inferior to healthy controls at Day 42, while rigorously quantifying common and serious adverse events. Secondary analyses explore viremia kinetics, T-cell immunity, antibody durability to one year, and host- or treatment-related modifiers of vaccine response.

By integrating comprehensive immunologic endpoints with robust safety monitoring, this trial will provide the first high-quality evidence to inform dengue vaccination policy for children, adolescents and adults living with ARDs in endemic regions-potentially broadening individual protection and supporting public-health efforts to mitigate dengue's impact in Brazil and similar settings.

ELIGIBILITY:
Inclusion Criteria:

* Age between 12 and 59 years
* Male or female
* Clinical diagnosis of an autoimmune rheumatic disease (ARD) based on internationally accepted criteria (e.g., rheumatoid arthritis, systemic lupus erythematosus, juvenile idiopathic arthritis, Sjögren's syndrome, vasculitis)
* Healthy control matched by age and sex
* ARD patients with clinically stable disease for at least 3 months
* ARD patients under low-grade immunosuppression or no immunosuppression
* Acceptable immunosuppressive treatments include:

Hydroxychloroquine Sulfasalazine Prednisone ≤ 20 mg/day Methotrexate ≤ 0.4 mg/kg/week (maximum 20 mg/week) Leflunomide 20 mg/day Azathioprine < 3 mg/kg/day Combination therapy with low-dose prednisone (≤ 7.5 mg/day), hydroxychloroquine, or sulfasalazine

* Healthy controls with no history of autoimmune or chronic infectious diseases
* Healthy controls not taking immunosuppressive medications Willing and able to comply with study procedures and follow-up
* Female participants of reproductive potential with negative pregnancy test at baseline
* Female participants of reproductive potential agreeing to use effective contraception for at least 90 days after vaccination

Exclusion Criteria:

* Prior receipt of any dengue vaccine
* Receipt of a live attenuated vaccine within 4 weeks prior to enrollment
* Receipt of an inactivated vaccine within 2 weeks prior to enrollment
* Known allergy to any component of the vaccine
* Febrile illness (≥ 37.8°C) within 72 hours prior to vaccination
* History of immunodeficiency syndromes
* History of asplenia
* History of cancer
* History of HIV infection
* History of primary immunodeficiencies
* Immunosuppression due to organ transplant
* Chronic uncontrolled comorbidities (e.g., heart failure, renal failure, hepatic insufficiency, diabetes mellitus)
* Hospitalization or acute illness at screening
* Receipt of blood transfusion within 3 months prior to enrollment
* Current pregnancy or breastfeeding
* Intention to become pregnant within 90 days post-vaccination
* Participation in another clinical trial within 30 days prior to enrollment

Ages: 12 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 477 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Seroconversion Rate After Vaccination | From enrollment to day 42 after vaccination
  Proportion of participants who achieve seroconversion (defined by PRNT50 neutralizing antibody titers) for any dengue serotype at Day 42 following a single dose of the Butantan-DV vaccine. Comparisons will be made between patients with autoimmune rheumatic diseases (ARDs) and healthy controls.
Frequency and Intensity of Common Adverse Events | Baseline through Day 42.
  Frequency and intensity of solicited local and systemic adverse events (e.g., pain at injection site, fever, headache, fatigue) with frequency up to 1/100, up to Day 42 post-vaccination, classified according to severity grading. Comparisons will be made between ARD patients and healthy controls.

SECONDARY OUTCOMES:
Disease Activity Flares After Vaccination | Day 1 to Day 42
  Number of patients with autoimmune rheumatic diseases (ARDs) who experience a flare or increase in disease activity, as defined by validated disease-specific indices (e.g., DAS28, SLEDAI-2K, ASDAS), between Day 1 and Day 42.
Frequency of Serious Adverse Events (SAEs) | Day 1 through Day 400
  To evaluate safety of the vaccine. Frequency of serious adverse events (hospitalizations, death, confirmed dengue with warning signs or severe dengue) occurring at any time during the study period in ARD patients compared to healthy controls.
Frequency of Adverse Events of Special Interest (AESIs) | Day 1 through Day 400
  Frequency of AESIs, including immune-mediated disorders, dengue infection post-vaccination, and other medically significant events, throughout the study duration.
Intensity of Viremia Post-Vaccination | Days 1, 7, 14, 28, 42, and 68 (if viremia is detected)
  Quantification and comparison of dengue viremia levels among ARD patients and healthy controls in a viremia substudy group, using RT-PCR at specified time points.
Duration of Viremia Post-Vaccination | Days 1, 7, 14, 28, 42, and 68 (if viremia is detected)
  Quantification, comparison and duration of dengue viremia levels among ARD patients and healthy controls in a viremia substudy group, using RT-PCR at specified time points.
Frequency of Grade 3 or 4 Adverse Events | Day 1 to Day 42
  Comparison of the frequency of grade 3 or 4 adverse events (as defined by severity scales) between ARD patients and healthy controls.
Geometric Mean Titers Against Dengue Serotypes | Day 1 and Day 42
  Comparison of the geometric mean antibody titers (GMTs) against DENV-1, DENV-2, DENV-3, and DENV-4 between ARD patients and healthy controls, as measured by PRNT50.
Factors Associated With Vaccine Immunogenicity | Day 1 and Day 42
  Identification of clinical and demographic variables associated with vaccine-induced antibody response in ARD patients, including prior dengue exposure, disease activity, and treatment regimen.
Persistence of Antibody Response | Day 400
  Evaluation of antibody titers against all four dengue serotypes one year post-vaccination in ARD patients and healthy controls.
Influence of Physical Activity Levels on Vaccine-Induced Humoral Immune Response | Day 1 to 14
  To assess the association between accelerometry-derived metrics (moderate-to-vigorous activity time, sedentary behavior, vector magnitude) and humoral immune response
Influence of dietary intake on Vaccine-Induced Humoral Immune Response | Day 1
  Dietary intake will be assessed using three non-consecutive 24-hour recalls, including one weekend day, analyzed via Dietbox software. Energy and macronutrient intake will be calculated, and food quality assessed based on the NOVA classification by level of processing.

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Hospital das Clínicas da Faculdade de Medicina da USP, São Paulo, São Paulo
  - Rheumatology Division, Faculdade de Medicina da USP, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thomas SJ, Yoon IK. A review of Dengvaxia(R): development to deployment. Hum Vaccin Immunother. 2019;15(10):2295-2314. doi: 10.1080/21645515.2019.1658503. Epub 2019 Oct 7. PMID 31589551
- [Background] Fernandez-Martinez S, Cortes X, Borras-Blasco J, Gracia-Perez A, Castera ME. Effectiveness of a systematic vaccination program in patients with autoimmune inflammatory disease treated with anti-TNF alpha drugs. Expert Opin Biol Ther. 2016 Nov;16(11):1317-1322. doi: 10.1080/14712598.2016.1218844. Epub 2016 Aug 18. PMID 27537179
- [Background] Biswal S, Reynales H, Saez-Llorens X, Lopez P, Borja-Tabora C, Kosalaraksa P, Sirivichayakul C, Watanaveeradej V, Rivera L, Espinoza F, Fernando L, Dietze R, Luz K, Venancio da Cunha R, Jimeno J, Lopez-Medina E, Borkowski A, Brose M, Rauscher M, LeFevre I, Bizjajeva S, Bravo L, Wallace D; TIDES Study Group. Efficacy of a Tetravalent Dengue Vaccine in Healthy Children and Adolescents. N Engl J Med. 2019 Nov 21;381(21):2009-2019. doi: 10.1056/NEJMoa1903869. Epub 2019 Nov 6. PMID 31693803
- [Background] Kallas EG, Cintra MAT, Moreira JA, Patino EG, Braga PE, Tenorio JCV, Infante V, Palacios R, de Lacerda MVG, Batista Pereira D, da Fonseca AJ, Gurgel RQ, Coelho IC, Fontes CJF, Marques ETA, Romero GAS, Teixeira MM, Siqueira AM, Barral AMP, Boaventura VS, Ramos F, Elias Junior E, Cassio de Moraes J, Covas DT, Kalil J, Precioso AR, Whitehead SS, Esteves-Jaramillo A, Shekar T, Lee JJ, Macey J, Kelner SG, Coller BG, Boulos FC, Nogueira ML. Live, Attenuated, Tetravalent Butantan-Dengue Vaccine in Children and Adults. N Engl J Med. 2024 Feb 1;390(5):397-408. doi: 10.1056/NEJMoa2301790. PMID 38294972